CLINICAL TRIAL: NCT06927531
Title: Effects of Pilates Ball and Sacral Massage Applications on Labor Pain, Labor Duration and Childbirth Satisfaction: A Randomized Controlled Study
Brief Title: Effects of Pilates Ball and Sacral Massage Applications on Labor Pain, Labor Duration and Childbirth Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, emine can, res. asst., Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Decision No: 24-9.1T/46
Record Dates: First submitted 2025-02-20; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Labor Pain; Satisfaction
Keywords: sacral massage; pilates ball
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sacral massage (Experimental): During labor, pregnant women will be given effleurage (stroking) and vibration (vibration) techniques to the sacral region in a comfortable position during contractions, once an hour for a maximum of 10 minutes.
  Interventions: Other: sacral massage
- pilates ball (Experimental): During labor, pregnant women will be made to perform pelvic oscillation movements (full rotation of the hips, going right/left, coming forward and back, gently bouncing on a ball while holding on to the headboard) once an hour during the active phase of labor.
  Interventions: Other: pilates ball
- control (No Intervention): Pregnant women in the control group will not be subjected to any intervention other than the routine practices of the clinic.

INTERVENTIONS:
Other: sacral massage — During labor, pregnant women will be given effleurage (stroking) and vibration (vibration) techniques to the sacral region in a comfortable position during contractions, once an hour for a maximum of 10 minutes.
  Arms: sacral massage
Other: pilates ball — During labor, pregnant women will be given pelvic oscillation movements (a full rotation of the hips, going right/left, coming forward and backward, lightly bouncing on a ball while holding onto the headboard) once an hour during the active phase of labor.
  Arms: pilates ball

SUMMARY:
As researchers, we believe that Pilates ball and manual sacral massage applications can be easily and cost-free applied in maternity clinics in our country. For all these reasons, this study was planned as a randomized controlled study to evaluate the effects of Pilates ball and sacral massage applications in labor on labor pain, labor duration, and labor satisfaction.

The research will be carried out between December 1, 2024 and May 1, 2025 in two public hospitals affiliated with the Gaziantep Provincial Health Directorate. The sample of the research will consist of 35 pregnant women in the Pilates ball group, 35 in the sacral massage group and 35 in the control group, totaling 105 pregnant women who meet the criteria for inclusion in the research. Applications to the intervention groups will be made during the active phase of labor. Personal Information Form, Labor Monitoring Form, Application Monitoring Form to record the number and duration of applications, Visual Analog Scale to assess labor pain, Partograph to assess labor duration and Labor Satisfaction Scale to assess maternal satisfaction will be used in data collection. Data will be analyzed with tests appropriate to normal distribution characteristics in the SPSS 24 package program. At the end of the research, the effects of Pilates ball and sacral massage applications in labor on labor pain, labor duration and labor satisfaction will be evaluated.

DETAILED DESCRIPTION:
Childbirth is one of the most special processes experienced in women's lives, significantly affecting their quality of life. Pain and fear experienced during the birth process are associated with many negative outcomes affecting the woman and the fetus/newborn, such as decreased childbirth satisfaction, preference for cesarean section, prolonged and difficult labor, and postpartum depression. Non-pharmacological methods that can be used to cope with labor pain are comfortable, safe, easy-to-use, and low-cost non-invasive methods that midwives can perform independently and in collaboration with the pregnant woman. Midwives working in delivery rooms should be able to apply non-pharmacological methods to cope with labor pain and should help teach and implement these methods by knowing their limitations and effects.

As researchers, we believe that Pilates ball and manual sacral massage applications can be easily and cost-free applied in maternity clinics in our country. For all these reasons, this study was planned as a randomized controlled study to evaluate the effects of Pilates ball and sacral massage applications in labor on labor pain, labor duration, and labor satisfaction.

The research will be carried out between December 1, 2024 and May 1, 2025 in two public hospitals affiliated with the Gaziantep Provincial Health Directorate. The sample of the research will consist of 35 pregnant women in the Pilates ball group, 35 in the sacral massage group and 35 in the control group, totaling 105 pregnant women who meet the criteria for inclusion in the research. Applications to the intervention groups will be made during the active phase of labor. Personal Information Form, Labor Monitoring Form, Application Monitoring Form to record the number and duration of applications, Visual Analog Scale to assess labor pain, Partograph to assess labor duration and Labor Satisfaction Scale to assess maternal satisfaction will be used in data collection. Data will be analyzed with tests appropriate to normal distribution characteristics in the SPSS 24 package program. At the end of the research, the effects of Pilates ball and sacral massage applications in labor on labor pain, labor duration and labor satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years old and under 35 years old
* Term pregnancies (38-41 weeks gestation)
* Primiparous
* Those with a single live fetus
* Vertex development
* Those who do not have any risk factors during pregnancy (Dermatological disease, Preeclampsia, active membrane rupture, oligohydramnios and polyhydramnios, gestational diabetes, placental anomalies, intrauterine growth retardation, intrauterine dead fetus, macrosomic babies, fetal distress, etc.)
* Those who do not have any obstacles for Pilates ball application
* Those who do not have any chronic diseases (Hypertension, DM, ...)
* Those in the active phase of labor, those who have at least 1 hour of labor follow-up
* Pregnant women who voluntarily accept to participate in the study

Exclusion Criteria:

* Indications for Caesarean section (such as presentation disorder, breech presentation)
* Those who underwent induction
* Those whose labor duration was shorter than 1 hour or longer than 8 hours
* Those who underwent vacuum forceps or shoulder insertion

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 105 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The intensity of pain will be measured with a visual pain scale. | prebirth during
  reduction in pain in intervention groups

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Unıversity, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makvandi S, Hadizadeh-Talasaz Z, Nosrati Hadi Abad SF, Manouchehri E, Larki M. Effectiveness of sacral massage during labor in pregnant women: A systematic review and meta-analysis. Midwifery. 2025 Feb;141:104252. doi: 10.1016/j.midw.2024.104252. Epub 2024 Nov 28. PMID 39673988
- [Background] https://doi.org/10.1111/jjns.12580
- [Background] Erkal Aksoy Y, Dereli Yilmaz S, Celimli S. Effect of using a birth ball on birth satisfaction and pain in pregnant women during labor: a randomized controlled trial. Arch Gynecol Obstet. 2024 Dec;310(6):2999-3007. doi: 10.1007/s00404-024-07825-3. Epub 2024 Nov 25. PMID 39585392